CLINICAL TRIAL: NCT05138887
Title: Clinical Professor
Brief Title: A Study for Assessing the Efficacy and Safety of BH4 in Radiation Enteritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, Clinical Professor, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCSUH2021001
Record Dates: First submitted 2021-10-11; First posted 2021-12-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Radiation Enteritis
Keywords: Tetrahydrobiopterin; Radiation Enteritis; Gynecological Cancer
MeSH Terms: interventions — sapropterin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo group (Placebo Comparator): The placebo group was administered a vitamin tablet (Centrum) orally, once a day
  Interventions: Drug: Tetrahydrobiopterin
- experimental group 1 (Experimental): The experimental group 1 was administered BH4 orally, with a dose of 2mg/kg.d (If the drug dose is within the range of 51-150mg, the drug dose will be 100mg), once per day
  Interventions: Drug: Tetrahydrobiopterin
- experimental group 2 (Experimental): The experimental group 2 was administered BH4 orally, with a dose of 5 mg/kg.d (If the drug dose is within the range of 151-250mg, the drug dose will be 200mg, two times a day; If the drug dose is within the range of 251-350mg, the drug dose will be 300mg, three times a day)
  Interventions: Drug: Tetrahydrobiopterin

INTERVENTIONS:
Drug: Tetrahydrobiopterin — The experimental group1 was administered BH4 orally with a dose of 2 mg/kg.d, once per day, and the experimental group 2 was administered BH4 orally witha dose of 5 mg/kg.d, two times a day (If the drug dose is within the range of 151-250mg, the drug dose is 200mg) or three times a day (If the drug dose is within the range of 251-350mg, the drug dose is 300mg). The oral administration of pills was started on the same day of the first radiation treatment, and ended three months after the treatment ended.

SUMMARY:
This present study envisaged a single-center, prospective, open-label, placebo and randomized controlled phase II clinical study to assess the efficacy and Safety of Tetrahydrobiopterin in Treating Radiation Enteritis in Gynecological Cancer Patients.

DETAILED DESCRIPTION:
Radiotherapy is one of the most effective treatments for pelvic malignancies. About 35~61% of the patients with pelvic cancer receive pelvic radiotherapy. Although radiotherapy significantly prolongs the survival time of the patients, it induces an injury to the normal tissues that may damage the pelvic and abdominal organs, with rectal damage as the most common and persistent adverse effect. Radiation proctitis refers to the rectal damage as a result of radiotherapy for the treatment of pelvic cancer such as cervical cancer, endometrial cancer, ovarian cancer, prostate cancer, rectal cancer, and bladder cancer. According to the time of onset and changing course of the disease, it can be divided into acute radiation-induced proctitis (ARP) and chronic radiation-induced proctitis (CRP), usually taking three months as a threshold. More than 75% of the patients receiving pelvic radiotherapy develop ARP, and 5%-20% of the patients develop CRP. In fact, the incidence of CRP is highly likely to be underestimated, since not every patient with symptoms goes for a clinical intervention. Studies have shown that 81% of the patients receiving pelvic radiotherapy developed gastrointestinal symptoms, but only 55% consulted the healthcare professionals. Approximately 90 % of the CRP patients exhibited permanent bowel habit changes, and 50% of the patients developed various gastrointestinal symptoms affecting their quality of life. Radiation enteritis seriously affects the treatment process of the patients, worsens the prognosis, and impairs the quality of life. The current common treatments for radiation enteritis are psychological intervention, anti-inflammatory drugs, antibiotics, probiotics to rebalance the gut microbiome, antioxidants, antidiarrheal agents, and surgical treatment, if necessary. However, the overall treatment effect does not yield satisfactory results. It is particularly important to find safe and effective preventive and treatment measures for the radiation enteritis to improve the prognosis of patients, and improve the quality of life.

Free radicals produced by the indirect action of ionizing radiation are considered to be one of the main causes of radiation enteritis. Tetrahydrobiopterin (BH4), also known as Sapropterin, is an important cofactor of the nitric oxide synthase (NOS) enzyme. Under normal physiological conditions, guanosine triphosphate cyclohydrolase 1 (GCH1) is the key enzyme for the synthesis of BH4. Reduction in GCH1 activity lowers the production of BH4, causes NOS uncoupling, and leads to an elevated level of oxygen free radicals (reactive oxygen species, ROS). Studies have shown that GCH1 over expression can restore BH4 level and NO products in irradiated skin cells, reverse and inhibit the NOS uncoupling caused by ionizing radiation, thereby eliminating the ionizing radiation-induced ROS, reducing DNA damage, and postponing the cell apoptosis and cell aging. In animal experiments, BH4 administration significantly reduced the occurrence of acute radiation enteritis.

This present study envisaged a single-center, prospective, open-label, placebo and randomized controlled phase II clinical study. The research subjects included the patients, who received radical radiotherapy and chemotherapy, and patients who needed supplementary radiotherapy due to prognostic risk factors for treating pathologically diagnosed gynecological malignancies (including cervical cancer, endometrial cancer, and vulvar cancer), with no pathological type restrictions.

The enrolled cases were randomly divided into three groups ina ratio of 1:1:1. The placebo group was administered a vitamin tablet (Centrum) orally, once a day. The two experimental groups were administered BH4 orally, with a dose of 100 mg, once per day, and a dose of 100 mg, three times a day (morning, noon, and evening). The oral administration of pills was started on the same day of the first radiation treatment, and ended three months after the treatment ended. The degree of injury of the radiation enteritis among the patients was evaluated weekly after the treatment started. It was evaluated one month and three months after the end of treatment, once per three months for two years and once per six months between 2~5 years after the treatment ended. The degree of ARP and CRP was evaluated according to the radiation morbidity scoring criteria of the Radiation Therapy Oncology Group (RTOG).

Intensity-modulated radiation therapy (IMRT) was adopted, using the conventional split mode,(1.8~2.0) Gy/day, 5 times/week.The pelvic clinical target volume (CTV) was(45~50.4)Gy/25~28 times, and the boost for local lymph nodes metastasis was raised to (60~70) Gy. Patients with indications for brachytherapy were treated with brachytherapy following the International Commission on Radiation Units & Measurements (ICRU) Report No. 89. The radical therapy treated or postoperative high-risk patients receiveda concurrent radiotherapy and chemotherapy, usingunrestricted chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18years old female patients.
2. Patients who received radical radiotherapy and chemotherapy, and who needed supplementary radiotherapy due to the prognostic risk factors for treating pathologically diagnosed gynecological malignancies (including cervical cancer, endometrial cancer, and vulvar cancer), with no pathological type restrictions.
3. The Eastern Cooperative Oncology GroupPerformance Status (ECOG PS) score: 0-1.
4. Expected survival ≥12 months.
5. The main organs functioned normally, which meant that they met the following criteria: Hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC)≥1.5×109/L; Platelet count (PLT) ≥50×109/L; Total bilirubin (TBIL)<1.5×upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<2.5×ULN,for patients with liver metastasis<5×ULN; Blood urea nitrogen (BUN) and Creatinine ratio (CR) ≤1×ULN or Endogenous creatinine clearance≥50ml/min(by Cockcroft-Gault equation).
6. The subjects willingly participated inthe study, signed an informed consent form, were medication-compliant, and cooperated with the follow-ups.

Exclusion Criteria:

1. Patients with hypertension and could not control the blood pressure within the normal range after treating with antihypertensive medications (systolic blood pressure>140 mmHg and diastolic blood pressure>90 mmHg).
2. Patients with a history of severe cardiovascular diseases, including myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (QTc interval ≥470 ms in women), grade III~IV cardiac insufficiencyaccording to the New York Heart Association (NYHA) standards, orthe left ventricular ejection fraction (LVEF) < 50%shown by the heart color Doppler ultrasound.
3. Patients with coagulation disorders (international normalized ratio (INR) >1.5, activated partial thromboplastin time (aPTT) >1.5 ULN), with bleeding tendency.
4. Patients with a history of psychotropic medication abuse and unable to quit, and patients with mental disorders.
5. Patients participatingin another drug trial.
6. Patients with concomitant diseases that seriously endangered the safety of the patient or affected the completion of the study from the investigators' opinion.
7. Not suitable for enrollment in the investigators' opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
acute radiation-induced proctitis (ARP) incidence | up to 12 weeks
  evaluated every week (according to RTOG radiation morbidity scoring criteria)

SECONDARY OUTCOMES:
chronic radiation-induced proctitis (CRP) incidence | up to 5 years
  according to RTOG radiation morbidity scoring criteria
progression-free survival (PFS) | up to 5 years
  Follow-up until the patient dies or withdraws from the study
overall survival (OS | up to 5 years
  Follow-up until the patient dies or withdraws from the study
cancer remission rate assessed by imaging | up to 12 weeks
  Until the end of treatment, The objective tumor response rate is used as the evaluation standard, which is divided into CR, PR, SD and PD

OTHER OUTCOMES:
quality of life (QoL) | up to 5 years
  Until the end of treatment, The quality of life assessment was performed using QLQ-C30 and QLQ-CX24, before treatment and at 3, 6, 9, and 12 months after treatment. results from multiple questionnaires will be reported.
adverse events | up to 5 years
  Follow-up until the patient dies or withdraws from the study

CONTACTS AND LOCATIONS:
Locations (1):
- est China Second Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng Y, Feng Y, Gu L, Liu P, Cao J, Zhang S. The Critical Role of Tetrahydrobiopterin (BH4) Metabolism in Modulating Radiosensitivity: BH4/NOS Axis as an Angel or a Devil. Front Oncol. 2021 Aug 27;11:720632. doi: 10.3389/fonc.2021.720632. eCollection 2021. PMID 34513700
- [Result] Thabet NM, Rashed ER, Abdel-Rafei MK, Moustafa EM. Modulation of the Nitric Oxide/BH4 Pathway Protects Against Irradiation-Induced Neuronal Damage. Neurochem Res. 2021 Jul;46(7):1641-1658. doi: 10.1007/s11064-021-03306-0. Epub 2021 Mar 23. PMID 33755856
- [Result] Yan T, Guo S, Zhang T, Zhang Z, Liu A, Zhang S, Xu Y, Qi Y, Zhao W, Wang Q, Shi L, Liu L. Ligustilide Prevents Radiation Enteritis by Targeting Gch1/BH4/eNOS to Improve Intestinal Ischemia. Front Pharmacol. 2021 Apr 22;12:629125. doi: 10.3389/fphar.2021.629125. eCollection 2021. PMID 33967762
- [Result] Xue J, Yu C, Sheng W, Zhu W, Luo J, Zhang Q, Yang H, Cao H, Wang W, Zhou J, Wu J, Cao P, Chen M, Ding WQ, Cao J, Zhang S. The Nrf2/GCH1/BH4 Axis Ameliorates Radiation-Induced Skin Injury by Modulating the ROS Cascade. J Invest Dermatol. 2017 Oct;137(10):2059-2068. doi: 10.1016/j.jid.2017.05.019. Epub 2017 Jun 6. PMID 28596000